CLINICAL TRIAL: NCT00790972
Title: The Efficacy of SinoFresh Nasal and Sinus Care Nasal Spray in Eliminating MRSA From the Nasal Cavity
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Company went out of business.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15419A
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: MRSA Infection
Keywords: MRSA; sinofresh; nasal spray

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator): Identical-appearing placebo
  Interventions: Drug: Placebo
- 1 (Active Comparator): two sprays in each nostril three times daily for one week
  Interventions: Drug: Sinofresh

INTERVENTIONS:
Drug: Sinofresh — two sprays in each nostril three times daily for one week
  Arms: 1
Drug: Placebo — two sprays in each nostril three times daily for one week
  Arms: 2

SUMMARY:
This is a study to assess the ability of SinoFresh Nasal & Sinus Care, an FDA approved over-the-counter nasal spray, to eliminate the bacteria in your nose.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* The volunteer is able to adhere to the study requirements and study visits.
* Agrees to abstain from use of other nasal sprays for length of study.
* Diagnosis of an MRSA carrier by PCR testing

Exclusion Criteria:

* History of chronic nose bleeds.
* History of intranasal steroids in the last 2 months
* Nasal obstruction severe enough to prohibit effective delivery of a nasal spray
* Epistaxis
* Significant excoriation in the opinion of the Investigator.
* Known hypersensitivity to any ingredients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2010-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
This is a study to assess the ability of SinoFresh Nasal & Sinus Care, an FDA approved over-the-counter nasal spray, to eliminate the bacteria in your nose. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Irsk Anderson, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States